CLINICAL TRIAL: NCT05143099
Title: Phase II Clinical Study on the Efficacy and Safety of Immune Checkpoint Inhibitor Combined With Cetuximab and Irinotecan in the Treatment of Recurrent, Refractory and Metastatic Colorectal Cancer
Brief Title: Phase II Study of Tislelizumab Combined With Cetuximab and Irinotecan in the Treatment of Recurrent, Refractory mCRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Director of Oncology Department, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEC
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): tislelizumab combined with cetuximab and irinotecan
  Interventions: Drug: TEC

INTERVENTIONS:
Drug: TEC — tislelizumab（an anti-PD-1 monoclonal antibody）+cetuximab（monoclonal antibody against EGFR）+irinotecan

SUMMARY:
This is a single arm, open phase II study to evaluate the efficacy and safety of tislelizumab combined with cetuximab + irinotecan in the treatment of Ras wild-type recurrent and refractory colorectal cancer. This study will include Ras wild-type colorectal cancer that failed at least second-line treatment in the past, including chemotherapy (oxaliplatin, irinotecan, fluorouracil) with or without targeted drugs (cetuximab, bevacizumab). 33 patients were planned to be treated with tislelizumab combined with cetuximab + irinotecan every 2 weeks. The enrollment time is expected to be 12 months and the follow-up is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years；
2. The ECOG PS score of the eastern United States cancer cooperation group was 0 or 1;
3. Ras wild-type colorectal cancer diagnosed by histology and / or cytology has metastasis or recurrence that cannot be cured by surgery;
4. Have received at least second-line systemic anti-tumor treatment for MCRC and failed, in which chemotherapy drugs can include fluorouracil, oxaliplatin and irinotecan, such as XELOX, FOLFOX, FOLFIRI, folfoxiri and xeliri; targeted drugs can be combined or not, such as cetuximab and bevacizumab;
5. At least one measurable lesion defined according to RECIST version 1.1;
6. Patients with fertility must be willing to take efficient contraceptive measures during the study period and ≥ 120 days after the last administration of tirelizumab; female patients have negative urine or serum pregnancy test results ≤ 7 days before the first administration of the study drug;
7. Fully understand this study and voluntarily sign the informed consent form.

Exclusion Criteria:

1. The following laboratory indicators belong to the exclusion criteria:

   1. Absolute neutrophil count (ANC) < 1.5 × 109 / L, or platelet count < 100 × 109 / L, or hemoglobin < 9g / dL or 90g / L or 5.6mmol/l; Blood transfusion or growth factor support within 2 weeks before enrollment are not allowed to meet the enrollment criteria;
   2. Serum total bilirubin > 1.5 times the upper limit of normal value (ULN); Patients with liver metastasis > 2.5 times ULN;
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5 times ULN, or ALT and / or ast > 5 times ULN in patients with liver metastasis;
   4. Serum creatinine > 1.5 times the upper limit of normal value (ULN), or creatinine clearance < 60ml / min (calculated according to Cockcroft Gault formula);
   5. Partial prothrombin time (APTT) or prothrombin time (PT) > 1.5 times ULN (subject to the normal value of clinical trial and Research Center);
   6. Albumin < 30g / L;
   7. Clinically significant electrolyte abnormalities;
2. Any previous histological or hematological ctDNA test showed mismatch repair gene deletion (dmmr), microsatellite instability (MSI-H) and BRAF mutant patients;
3. Previous immunotherapy, including anti-PD-1, anti-PD-L1, anti-CTLA-4 or any cellular immunotherapy;
4. Have a history of active autoimmune disease or autoimmune disease that may recur;
5. Patients with any disease requiring systemic treatment with corticosteroids (the dose of prednisone or equivalent drug > 10 mg / day) or other immunosuppressive drugs within ≤ 14 days before the administration of the first study drug need not be excluded if they have used any of the following steroid treatment schemes at present or in the past:

   1. Adrenal replacement steroids (dose of prednisone or equivalent ≤ 10 mg / day);
   2. Local, ocular, intra-articular, intranasal or inhaled corticosteroids with very low systemic absorption;
   3. Short term (≤ 7 days) prophylactic use of corticosteroids (e.g. for the treatment of contrast medium allergy) or for the treatment of non autoimmune diseases (e.g. delayed type hypersensitivity caused by contact allergens);
6. there are a history of interstitial lung disease, non infectious pneumonia, pulmonary fibrosis, acute lung disease, or poorly controlled systemic diseases (including but not limited to diabetes, hypertension, etc.).
7. Clinically uncontrollable diarrhea;
8. chronic or active infections require systemic antibacterial, antifungal or antiviral treatment, including tuberculosis infection. Patients with a history of active tuberculosis infection ≥ 1 year before screening should also be excluded, unless proof can be provided that appropriate treatment has been completed;
9. Brain metastasis or leptomeningeal metastasis;
10. Clinically significant pleural effusion, pericardial effusion or ascites need to be drained for many times within 2 weeks before the first administration of the study drug;
11. There is a clinically detectable second primary malignant tumor at the time of enrollment, or there have been other malignant tumors in the past 5 years (except fully treated skin basal cell carcinoma or cervical carcinoma in situ);
12. despite the use of standard care, patients with poor control of diabetes or poor electrolyte control are still in control.
13. Known history of human immunodeficiency virus infection;
14. Untreated patients with chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA higher than 500 IU / ml and patients with positive hepatitis C virus (HCV) RNA should be excluded. Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA < 500 IU / ml), and cured hepatitis C patients were all selected;
15. Any major surgical operation ≤ 28 days before the administration of the first study drug;
16. Previous allogeneic stem cell transplantation or organ transplantation;
17. Uncontrollable hypertension, i.e. systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg after single drug treatment;
18. At present, there are gastrointestinal diseases such as duodenal ulcer, ulcerative colitis and intestinal obstruction, or other conditions that may cause gastrointestinal bleeding or perforation determined by the researchers; Or those who have a history of intestinal perforation and intestinal fistula and are not cured after surgical treatment;
19. Patients with a history of arterial thrombosis or deep venous thrombosis within 6 months before enrollment, or with evidence or history of bleeding tendency within 2 months before enrollment, regardless of severity;
20. Stroke or transient ischemic attack occurred within 12 months before enrollment;
21. Skin wound, operation site, wound site, severe mucosal ulcer or fracture are not fully healed;
22. Acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; Or patients with cardiac insufficiency of NYHA grade 2 or above;
23. Severe hypersensitivity to other monoclonal antibodies, irinotecan and its excipients;
24. Have received any systemic chemotherapy within 28 days before the first study drug, or received immunotherapy (such as interleukin, interferon, thymosin), hormone therapy, targeted therapy, or any research therapy within 14 days or 5 half lives before the first study drug, whichever is shorter;
25. Received any Chinese herbal medicine or proprietary Chinese medicine for cancer control within 14 days before the first study drug;
26. Patients whose toxic and side effects (due to previous anticancer treatment) have not returned to baseline or stable levels, unless it is not considered that such AE may pose safety risks (such as hair loss, neuropathy and specific laboratory abnormalities);
27. Have received live vaccine within 4 weeks (including) before the first administration of the study drug; Seasonal influenza vaccines are usually inactivated, so they are allowed to be used; Intranasal vaccine belongs to live vaccine, so it is not allowed to be used;
28. The investigator considers that the subject has any clinical or laboratory abnormalities or compliance problems and is not suitable to participate in this clinical study;
29. Serious psychological or mental abnormalities;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months after the last subject participating in
  proportion of patients with complete and partial remission in the best efficacy

SECONDARY OUTCOMES:
Disease control rate (DCR) | 24 months after the last subject participating in
  the best efficacy is the proportion of patients with complete remission, partial remission and stable disease
Progression free survival time (PFS） | 24 months after the last subject participating in
  time from the start of medication to the initial progression of the disease
Overall survival (OS） | 36 months after the last subject participating in
  time from the start of medication to death

OTHER OUTCOMES:
biomarker analysis | 12 months after the last subject participating in
  PD-L1 expression, tumor mutation burden (TMB) and proteins in blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Tianshu Liu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes